CLINICAL TRIAL: NCT06279663
Title: A Prospective Multicenter Randomized Trial: Management Tactics for Patients High Risk With Acute Coronary Syndrome Without ST Segment Elevation and Multivessel Coronary Artery Disease
Brief Title: Management Tactics for Patients High Risk With Acute Coronary Syndrome Without ST Segment Elevation and Multivessel Coronary Artery Disease
Acronym: NSTE-ACSMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Institution National Medical Research Center named after academician E.N. Me (Other Government)
Collaborators: Kemerovo Cardiology Center, Tarasov Roman Sergeevich (Unknown); Tomsk National Research Medical Center of the Russian Academy of Sciences, Ryabov Vyacheslav Valeryevich (Unknown)
Responsible Party: Principal Investigator, Obedinskiy Anton Andreyevich, Obedinskiy Anton Andreyevich, Federal State Budgetary Institution National Medical Research Center named after academician E.N. Me
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSTE-ACS Multivessel Trial
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Coronary Syndrome, Acute, Non-ST Elevation, High Risk Patients
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI (Active Comparator): complete revascularization
  Interventions: Procedure: Revascularization
- CABG (Active Comparator)
  Interventions: Procedure: Revascularization

INTERVENTIONS:
Procedure: Revascularization — revascularization

SUMMARY:
The study will include patients with acute coronary syndrome without ST segment elevation and multivessel CA lesion, who are subject to surgical treatment according to KG data (Syntax Score 23 - 32 points with significant damage to the anterior descending artery and/or trunk of the left coronary artery). The patient should be suitable for both CABG and PCI (confirmed by an X-ray surgeon and a cardiac surgeon). An X-ray surgeon and a cardiac surgeon, within the framework of planning the volume of revascularization, strives for the fullest feasible volume. Complete myocardial revascularization (that is, the desire for the absence of hemodynamically significant coronary arteries after revascularization, with a diameter of > 2.5 mm, that is, residual coronary artery stenosis of no more than 60%). Thus, patients will be randomized into groups in a ratio of 1:1. Each group will need to include 230 patients (a total of 460). In the main group, revascularization will be performed by PCI, in the control group by CABG.

ELIGIBILITY:
Inclusion Criteria:

1. Acute coronary syndrome without ST segment elevation of high risk: unstable angina pectoris or myocardial infarction requiring revascularization within 24 hours based on the risk of an unfavorable outcome (increase or decrease in the concentration of cardiac troponin in the blood that meet the criteria of MI; dynamic ST segment displacement or changes in T; risk on the GRACE scale >140 points)
2. The patient is suitable for both CABG and PCI, confirmed by an interventional cardiologist and surgeon (multivessel lesion with a Sintax score of 23-32 points with significant damage to the anterior descending artery and/or trunk of the left coronary artery).
3. Complete myocardial revascularization (that is, the desire for the absence of hemodynamically significant coronary arteries after revascularization, with a diameter of > 2.5 mm, that is, residual coronary artery stenosis of no more than 60%).
4. Signed informed consent
5. Age over 18 years.

Exclusion Criteria:

1. Myocardial infarction with ST segment elevation
2. Stable angina pectoris
3. Patients with OSN Killip II-IV class
4. Patients required an immediate PCI procedure (e.g. electrical instability)
5. A history of hemorrhagic stroke one year before the procedure
6. Ischemic stroke or TIA in the last 6 weeks
7. The final stage of chronic renal failure requiring dialysis.
8. Preliminary PCI for any other coronary artery lesion within 1 year prior to randomization.
9. Pre-CABG at any time prior to randomization.
10. The need for concomitant cardiac surgery, except for CABG (for example, valve surgery, aortic repair, etc.). Patients who require additional surgery (cardiological or extra-cardiac) for 1 year.
11. Non-cardiac concomitant diseases with a life expectancy of less than 1 year (for example, oncological diseases).

13. The left ventricular ejection fraction is less than 40%. 14. Severe degree of COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 460 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Death from any cause | 1 year
  a fatal outcome due to any cause or disease
Combined endpoint (death from cardiovascular causes, MI, Stroke, repeated unplanned myocardial revascularization) | 1 year
  Death from cardiovascular causes, MI, Stroke, repeated unplanned myocardial revascularization.
target LDL level | 1 year
  Achieved target LDL level

SECONDARY OUTCOMES:
Myocardial infarction | 1 year
  Myocardial infarction (Fourth universal definition of myocardial infarction (2018))
Stroke | 1 year
  clinically verified acute cerebrovascular accident of any etiology (hemorrhagic or ischemic)
Repeated unplanned myocardial revascularization | 1 year
  any type of repeated myocardial revascularization by endovascular or cardiac surgery performed in the time period after index revascularization;
Duration of the hospital period | 1 year
  the number of bed days that the patient spent in the clinic in connection with an index event and/or complications arising from the underlying, concomitant diseases, as well as in connection with the treatment.
Intra/perioperative complications | 1 year
  Any intra/perioperative complications (MI, Stroke, hemorrhagic complication, )
Significant hemorrhagic complications (grade 3 or more on the BARC scale) | 1 year
  any bleeding that occurred during or after the index revascularization of the myocardium, leading to a clinically significant decrease in hemoglobin levels, requiring hemotransfusion and/or surgical methods of hemostasis, artery dissection, shunt thrombosis, and other
Questionnaire | 1 year
  SF-36 Quality of Life Questionnaire and Rose Questionn

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Anton, Novosibirsk, Novosibirsk Obl
  - Anton, Novosibirsk, Rechkunovskaya Str.

IPD SHARING:
Plan to Share IPD: Undecided